CLINICAL TRIAL: NCT06665646
Title: A Phase 1 Open-label, Non-randomized, Clinical Trial to Evaluate the Safety and Immunogenicity of Hiltonol, Poly-ICLC-adjuvanted CD40.HIVRI.Env (VRIPRO) in Adult Participants Who Previously Participated in HVTN 706
Brief Title: Clinical Trial to Evaluate the Safety and Immunogenicity of Hiltonol, Poly-ICLC-adjuvanted CD40.HIVRI.Env (VRIPRO) in Adult Participants Who Previously Participated in HVTN 706
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 318
Record Dates: First submitted 2024-09-17; First posted 2024-10-30 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1- Study product received in HVTN 706: Study Vaccine (Experimental): Participants will receive Hiltonol, Poly-ICLC-adjuvanted CD40.HIVRI.Env(VRIPRO) as a subcutaneous injection.
  Interventions: Biological: CD40.HIVRI.Env (VRIPRO); Biological: Hiltonol Poly-ICLC-adjuvant
- Group 2 - Study product received in HVTN 706: Placebo (Experimental): Participants will receive Hiltonol, Poly-ICLC-adjuvanted CD40.HIVRI.Env(VRIPRO) as a subcutaneous injection.
  Interventions: Biological: CD40.HIVRI.Env (VRIPRO); Biological: Hiltonol Poly-ICLC-adjuvant

INTERVENTIONS:
Biological: CD40.HIVRI.Env (VRIPRO) — To be administered subcutaneously as 1 mg admixed with Hiltonol, Poly-ICLC as a single dose.
Biological: Hiltonol Poly-ICLC-adjuvant — Vaccine adjuvant

SUMMARY:
The clinical schedule will consist of 3 injections of CD40.HIVRI.Env (VRIPRO) at weeks 0, 4, and 24.40 volunteers without HIV and in overall good health, aged 18 to 60 years, who previously participated in the HVTN 706 trial.

ELIGIBILITY:
Inclusion Criteria:

1. Formerly participated in HVTN 706 study as active vaccine arm or placebo recipient (those enrolled in the active vaccine arm of HVTN 706 must have received all 4 vaccinations according to the HVTN 706 protocol).
2. Demonstrates an understanding of the study and is able and willing to complete the informed consent process.
3. 18 to ≤ 60 years old, on day of enrollment.
4. Available for clinic follow-up through the last clinic visit, willing to undergo FNA, and willing to be contacted 12 months after the last study-product administration.
5. Agrees not to enroll in another study of an investigational agent during participation in the trial. If a potential participant is already enrolled in another clinical trial, approvals from the other trial sponsor and the HVTN 318 (Protocol Safety Review Team) PSRT are required prior to enrollment into HVTN 318. Previous enrollment in HVTN 706 study is a requirement, per inclusion criteria 1.
6. In good general health according to the clinical judgment of the site investigator.
7. Physical examination and laboratory results without clinically significant findings that would interfere with assessment of safety or reactogenicity in the clinical judgement of the site investigator.
8. Agrees to discuss the potential for HIV acquisition and agrees to prevention counseling.
9. Hemoglobin (Hgb):

   * ≥11.0 g/dL for women
   * ≥13.0 g/dL for men
   * If receiving exogenous hormones for more than 6 consecutive months with dosing equivalent to parenteral testosterone ≥1000 mg every 12 weeks or estradiol valerate ≥2 mg/week, determine hemoglobin eligibility based on the exogenous hormone reported.
10. White blood cell (WBC) count = 2,500 to 12,000/mm^3 (WBC over 12,000/mm^3 is not exclusionary if further evaluation shows general good health and if PSRT approval is granted).
11. Platelets = 125,000 to 550,000/mm^3.
12. Alanine aminotransferase (ALT) < 2.5 x upper limit of institutional reference range.
13. Serum creatinine ≤ 1.1 x upper limit of normal (ULN) based on the institutional normal range.
14. Systolic blood pressure of 90 to < 140 mmHg and diastolic blood pressure of 50 to < 90 mmHg at screening visit. The average blood pressure between the screening visit and the enrollment visit must be below 140 mmHg systolic and 90 mmHg diastolic. A single measurement ≥ 160 systolic mmHg or 100 mmHg diastolic during the current study evaluation is exclusionary.
15. Negative HIV test results by one of the following options:

    * For participants who received study product under HVTN 706

      * A negative result from a HVTN HIV Diagnostic Testing Laboratory within 14 days prior to enrollment (see HVTN 318 HIV testing SSP for additional details); or
      * A negative result from a non-HVTN laboratory following the external guidance for non-HVTN laboratories within 14 days prior to enrollment (external laboratory guidance for non-HVTN laboratories can be found in the guidance document, HIV Infection and VISP/R Status Diagnostic Testing at External (non-HVTN Laboratories).
    * For participants at who received placebo under HVTN 706

      * A negative US Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA); or a chemiluminescent microparticle immunoassay (CMIA); or
      * A negative result on 2 different HIV rapid tests (one of these rapid tests must be FDA approved)
16. Negative for anti-Hepatitis C virus (HCV) Abs (anti-HCV) or negative HCV nucleic acid test (NAT) if anti-HCV antibodies (Abs) are detected.
17. Negative for Hepatitis B surface antigen (Ag).
18. Women with pregnancy potential:

    * Must have a negative β-HCG pregnancy test (urine or serum) on day of enrollment.
    * Must agree to use effective means of contraception from at least 21 days prior to enrollment until 8 weeks after their last scheduled vaccination. See Appendix D.
    * Women who have had a total hysterectomy, bilateral oophorectomy, or bilateral salpingectomy Consider including the cyan-highlighted parenthetical for product-specific reasons: (verified by medical records) or menopause (no menses for ≥1 year) are not required to undergo pregnancy testing.
19. Female volunteers must agree to not seek pregnancy through alternative methods, such as oocyte retrieval, artificial insemination, or in vitro fertilization from at least 21 days prior to enrollment through 8 weeks after their last scheduled vaccination timepoint.

Exclusion Criteria:

1. Body mass index (BMI) ≥ 40. Enrollment of individuals with BMI ≥ 40, whom the site investigator assesses are in good health, may be considered by PSRT approval.
2. Diabetes mellitus (DM). Type 2 DM controlled with diet alone (and confirmed by HgbA1c ≤ 8% within the last 6 months) or a history of isolated gestational diabetes are not exclusionary. Enrollment of individuals with Type 2 DM that is well controlled on hypoglycemic agent(s) may be considered by the PSRT on a case-by-case basis, provided that the HgbA1c is ≤ 8% within the last 6 months (sites may draw these at screening).
3. Previous or current recipient of an investigational HIV vaccine (not applicable to previous placebo/control recipients), with the exception of the HVTN 706 vaccine regimen as per Inclusion Criteria #1.
4. Receipt of non-HIV investigational vaccine(s) received within the last 1 year. Exceptions include vaccines that have subsequently undergone licensure or Emergency Use Authorization (EUA) by the FDA or World Health Organization (WHO) Emergency Use Listing (EUL), or if outside the US, by the national Regulatory Authority (RA) authorizing this clinical trial.
5. Congenital or acquired immunodeficiency, including systemic medication use likely to impair immune response to vaccine in the opinion of the site investigator, such as glucocorticoid use, ≥ prednisone 10 mg/day within 3 months prior to enrollment.
6. Blood products or immunoglobulin within 16 weeks prior to enrollment; receipt of immunoglobulin within 16 weeks prior to enrollment requires PSRT approval.
7. Receipt of any vaccine within 4 weeks prior to enrollment
8. Initiation of Ag-based immunotherapy for allergies within the previous year (stable immunotherapy is not exclusionary); inclusion of participants who initiated immunotherapy within the previous year requires PSRT approval.
9. Receipt of investigational research agents with a half-life of 7 or fewer days within 4 weeks prior to enrollment. If a potential participant has received investigational agents with a half-life of more than 7 days (or unknown half-life) within the past year, PSRT approval is required for enrollment.
10. Use of injectable long-acting Cabotegravir within 18 months prior to enrollment.
11. Serious adverse reactions to any vaccine, including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not applicable to a participant who had a non-anaphylactic adverse reaction to pertussis vaccine as a child.)
12. Hereditary angioedema, acquired angioedema, or idiopathic forms of angioedema.
13. Idiopathic urticaria within the past year.
14. Bleeding disorder diagnosed by a clinician that would make study procedures a contraindication.
15. History of seizure(s) within the past 3 years. Also applies to volunteer using medications in order to prevent or treat seizure(s) at any time within the past 3 years.
16. Asplenia or functional asplenia.
17. Active duty and reserve US military personnel.
18. Any other chronic or clinically significant condition that, in the clinical judgment of the investigator, would jeopardize the safety or rights of the study participant, including but not limited to: clinically significant forms of substance use or alcohol use disorder(s), serious psychiatric disorders, any suicide attempt within the past 1 year (if between 1 and 2 years, consult PSRT for approval), or cancer that, in the clinical judgement of the site investigator, has potential for recurrence (excluding basal cell carcinoma).
19. Asthma patients will not be enrolled if the volunteer has ANY of the following:

    * Required either oral or parenteral corticosteroids for an exacerbation 2 or more times within the past year; OR
    * Needed emergency care, urgent care, hospitalization, or intubation for an acute asthma exacerbation within the past year (eg, would NOT exclude individuals with asthma who meet all other criteria but sought urgent/emergent care solely for asthma medication refills or coexisting conditions unrelated to asthma); OR
    * Uses a short-acting rescue inhaler more than 2 days per week for acute asthma symptoms (ie, not for preventive treatment prior to athletic activity); OR
    * Uses medium- to high-dose inhaled corticosteroids (> 250 mcg fluticasone or therapeutic equivalent per day), whether in single-therapy or dual-therapy inhalers (ie, with a long-acting beta agonist [LABA]); OR
    * Uses more than 1 medication for maintenance therapy daily. Inclusion of anyone on a stable dose of more than 1 medication for maintenance therapy daily for greater than 2 years requires PSRT approval.
20. A participant with a history of a potential immune-mediated medical condition (PIMMC), either active or remote. Specific examples are listed in Appendix F (AESI Index). Not exclusionary: 1) Remote history of Bell's palsy (> 2 years ago) not associated with other neurologic symptoms and 2) mild psoriasis or other mild, uncomplicated, localized, or dermatologic condition that does not require ongoing systemic treatment.
21. History of allergy to local anesthetic (Novocaine, Lidocaine).
22. Volunteer who is breastfeeding or pregnant.
23. Investigator concern for difficulty with venous access based on clinical history and physical examination. For example, persons with a history of intravenous drug use or substantial difficulty with previous blood draws.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-14 (Actual); Primary Completion 2026-07-27 (Estimated); Study Completion 2027-05-04 (Estimated)

PRIMARY OUTCOMES:
Local signs and symptoms will be collected for a minimum of 14 days following receipt of adjuvanted CD40.HIVRI.Env (VRIPRO) | For a minimum of 14 days following receipt of adjuvanted CD40.HIVRI.Env (VRIPRO)
  Local events at the injection site include pain/tenderness, induration and erythema. These will be graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 (exceptions apply)
Systemic reactogenicity signs and symptoms will be collected | For a minimum of 14 days following receipt of adjuvanted CD40.HIVRI.Env (VRIPRO)
  Systemic events include increased body temperature, fatigue, generalized myalgia, generalized arthralgia, headache, chills, and nausea. These will be graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events,Corrected Version 2.1, July 2017 (exceptions apply)
Number of SAEs leading to early participant withdrawal or permanent discontinuation will be collected throughout the study and for 1 year following study product | 30 days after receipt of study vaccination up to 1 year following study product
Number of MAAEs leading to early participant withdrawal or permanent discontinuation will be collected throughout the study and for 1 year following study product | 30 days after receipt of study vaccination up to 1 year following study product
Number of AESIs leading to early participant withdrawal or permanent discontinuation will be collected throughout the study and for 1 year following study product | 30 days after receipt of study vaccination up to 1 year following study product
Number of AEs leading to early participant withdrawal or permanent discontinuation will be collected throughout the study and for 1 year following study product | 30 days after receipt of study vaccination up to 1 year following study product
Response rate of HIV-1-specific serum IgG binding antibodies against autologous and heterologous Env antigens as assessed by binding Ab multiplex assay (BAMA) in HVTN 706 regimen recipients | 2 weeks after receipt of the full CD40.HIVRI.Env (VRIPRO) regimen
Magnitude of HIV-1-specific serum IgG binding antibodies against autologous and heterologous Env antigens as assessed by binding Ab multiplex assay (BAMA) in HVTN 706 regimen recipients | 2 weeks after receipt of the full CD40.HIVRI.Env (VRIPRO) regimen
Response rate of HIV-1-specific serum IgG binding antibodies against autologous and heterologous V1V2 antigens as assessed by BAMA in HVTN 706 regimen recipients | 2 weeks after receipt of the full CD40.HIVRI.Env (VRIPRO) regimen
Magnitude of HIV-1-specific serum IgG binding antibodies against autologous and heterologous V1V2 antigens as assessed by BAMA in HVTN 706 regimen recipients | 2 weeks after receipt of the full CD40.HIVRI.Env (VRIPRO) regimen

SECONDARY OUTCOMES:
Response rate of serum HIV-1-specific IgG binding antibodies against autologous and heterologous Env antigens as assessed by binding Ab multiplex assay (BAMA) | 2 weeks after the receipt of the full CD40.HIVRI.Env (VRIPRO) regimen
Magnitude of serum HIV-1-specific IgG binding antibodies against autologous and heterologous Env antigens as assessed by binding Ab multiplex assay (BAMA) | 2 weeks after the receipt of the full CD40.HIVRI.Env (VRIPRO) regimen
Response rate of serum-HIV-1 specific IgG binding antibodies against autologous and heterologous V1V2 antigens as assessed by BAMA | 2 weeks after receipt of the full CD40.HIVRI.Env (VRIPRO) regimen
Magnitude of serum-HIV-1 specific IgG binding antibodies against autologous and heterologous V1V2 antigens as assessed by BAMA | 2 weeks after receipt of the full CD40.HIVRI.Env (VRIPRO) regimen
Response rate of serum HIV-1 specific IgG3 binding antibodies against autologous V1V2 antigens as assessed by BAMA | 2 weeks after receipt of the full CD40.HIVRI.Env (VRIPRO) regimen
Magnitude of serum HIV-1 specific IgG3 binding antibodies against autologous V1V2 antigens as assessed by BAMA | 2 weeks after receipt of the full CD40.HIVRI.Env (VRIPRO) regimen
Response rate of serum HIV-1 specific IgG3 binding antibodies against heterologous V1V2 antigens as assessed by BAMA | 2 weeks after receipt of the full CD40.HIVRI.Env (VRIPRO) regimen
Magnitude of serum HIV-1 specific IgG3 binding antibodies against heterologous V1V2 antigens as assessed by BAMA | 2 weeks after receipt of the full CD40.HIVRI.Env (VRIPRO) regimen
Response rate of serum Ab neutralization of autologous HIV-1 strains as measured by the TZM-bl assay | 2 weeks after receipt of the CD40.HIVRI.Env (VRIPRO) regimen
Magnitude of serum Ab neutralization of autologous HIV-1 strains as measured by the TZM-bl assay | 2 weeks after receipt of the CD40.HIVRI.Env (VRIPRO) regimen
Response rate of serum Ab neutralization of heterologous HIV-1 strains as measured by TZM-bl assay | 2 weeks after receipt of the CD40.HIVRI.Env (VRIPRO) regimen
Magnitude of serum Ab neutralization of heterologous HIV-1 strains as measured by TZM-bl assay | 2 weeks after receipt of the CD40.HIVRI.Env (VRIPRO) regimen
Response rate of CD4+ and CD8+ T-cell responses as assessed by intracellular cytokine staining, Epimax, or other assays, as needed | 2 weeks after receipt of the CD40.HIVRI.Env (VRIPRO) regimen
Magnitude of CD4+ and CD8+ T-cell responses as assessed by intracellular cytokine staining, Epimax, or other assays, as needed | 2 weeks after receipt of the CD40.HIVRI.Env (VRIPRO) regimen
Response rate of antibody-dependent cellular cytotoxicity (ADCC) | at baseline and 2 weeks after the last vaccination
Magnitude of antibody-dependent cellular cytotoxicity (ADCC) | at baseline and 2 weeks after the last vaccination
Response rate of antibody-dependent cellular phagocytosis (ADCP) | at baseline and 2 weeks after the last vaccination
Magnitude of antibody-dependent cellular phagocytosis (ADCP) | at baseline and 2 weeks after the last vaccination
Magnitude of Env-specific binding Abs assessed by the slope of BAMA titers | weeks 26 and 48
Frequency of total memory B cells and vaccine-specific B cell receptors | 2 weeks after receipt of the full CD40.HIVRI.Env (VRIPRO) regimen

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Bridge HIV CRS, San Francisco, California
  - The Hope Clinic of the Emory Vaccine Center CRS, Decatur, Georgia
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Columbia P&S CRS, New York, New York
  - Penn Prevention CRS (Site ID# 30310), Philadelphia, Pennsylvania
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No